CLINICAL TRIAL: NCT04665232
Title: Immunomodulatory Effects of Subcutaneous Progesterone in Patients Undergoing IVF Affected by Autoimmune Diseases
Brief Title: Immunomodulatory Effects of Subcutaneous Progesterone in Patients Affected by Autoimmune Diseases
Status: Completed | Type: Observational
Sponsor: San Carlo Public Hospital, Potenza, Italy (Other)
Responsible Party: Principal Investigator, Assunta Iuliano, MD, MD, PhD, San Carlo Public Hospital, Potenza, Italy
Other Study IDs: San Carlo Public Hospital
Record Dates: First submitted 2016-02-25; First posted 2020-12-11 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Autoimmune Diseases; Infertility
Keywords: autoimmune diseases and infertility; luteal supplementation with subcutaneous progesterone; Systemic effect of progesterone
MeSH Terms: conditions — Autoimmune Diseases; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients affected by autoimmune diseases: Infertile patients suffering from autoimmune diseases to be subjected to IVF in which the luteal phase has been supplemented with 25 mg /die of aqueous subcutaneous progesterone
  Interventions: Drug: aqueous subcutaneous progesterone

INTERVENTIONS:
Drug: aqueous subcutaneous progesterone — 25 mg/die of aqueous subcutaneous progesterone from the day of oocytes retrieval for two weeks.

SUMMARY:
This study evaluates the immunomodulatory effects of subcutaneous progesterone in patients undergoing IVF by determination of anti-nuclear antibodies (ANA),extractable nuclear antigen antibodies (ENA),anti- neutrophil cytoplasmic antibodies(ANCA),anti-DNA antibodies, anti-cardiolipin antibodies (ACA),Lupus anticoagulant antibodies (LAC) and C3 and C4 fractions of complement on the day of beta hCG dosage and during the eigth week of gestation.

DETAILED DESCRIPTION:
The aqueous progesterone preparation for s.c. injection is the first systemic progesterone of its kind for the provision of luteal phase support (LPS) in patients undergoing IVF.

The the high solubility and rapid absorption of the new preparation are enhanced using cyclodextrins that are starch residues with no therapeutic activity and with a particular molecular structure that closely resembles a 'cap'.

Once absorbed after injection, the progesterone molecule is immediately dissociated from its cyclodextrin 'cap', remaining free in the circulation as if produced endogenously by the ovaries.

In comparison to progesterone-in-oil preparation, the new aqueous solution administered by s.c.route resulted in a 3 fold higher and more rapid progesterone peak serum concentrations.

The immunomodulating effects of progesterone are mediated outside of the pelvic cavity, on the peripheral cell of the immune system. For this reason only the injection procedure has this advantage Furthermore, the faster absorption rate and the higher peak serum concentration should increas the systemic immunomodulatory effect of subcutaneous progesterone compared to the vaginal and intramuscular administration

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients affected by autoimmune diseases undergoing IVF

Exclusion Criteria:

* infertile patients without autoimmune diseases, fertile patients affected by autoimmune diseases

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile patients affected by autoimmune diseases undergoing IVF
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pregnancy Rate percentage, Implantation Rate percentage, Live Birth Rate percentage | 12 mounths
  number of pregnancies / 100 embryotransfer, number of implanted embryos/ number of embryos trafsferred, number of live birth

CONTACTS AND LOCATIONS:
Overall Officials: Assunta Iuliano, MD,PhD, Principal Investigator — San Carlo Public Hospital, Potenza, Italy
Locations (1):
- Assunta Iuliano, Potenza, Italy

IPD SHARING:
Plan to Share IPD: Yes
We have a register which shows the number of the medical record of the patient
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 30 years
Access Criteria: Archive of Medically Assisted Procreation of San Carlo Hospital

REFERENCES:
- [Background] Paulson RJ. Hormonal induction of endometrial receptivity. Fertil Steril. 2011 Sep;96(3):530-5. doi: 10.1016/j.fertnstert.2011.07.1097. PMID 21880274
- [Background] de Ziegler D, Sator M, Binelli D, Leuratti C, Cometti B, Bourgain C, Fu YS, Garhofer G. A randomized trial comparing the endometrial effects of daily subcutaneous administration of 25 mg and 50 mg progesterone in aqueous preparation. Fertil Steril. 2013 Sep;100(3):860-6. doi: 10.1016/j.fertnstert.2013.05.029. Epub 2013 Jun 24. PMID 23806850
- [Background] Practice Committee of the American Society for Reproductive Medicine. Current clinical irrelevance of luteal phase deficiency: a committee opinion. Fertil Steril. 2015 Apr;103(4):e27-32. doi: 10.1016/j.fertnstert.2014.12.128. Epub 2015 Feb 11. PMID 25681857
- [Background] Fatemi HM. The luteal phase after 3 decades of IVF: what do we know? Reprod Biomed Online. 2009;19 Suppl 4:4331. PMID 20034417
- [Background] Stavreus-Evers A, Mandelin E, Koistinen R, Aghajanova L, Hovatta O, Seppala M. Glycodelin is present in pinopodes of receptive-phase human endometrium and is associated with down-regulation of progesterone receptor B. Fertil Steril. 2006 Jun;85(6):1803-11. doi: 10.1016/j.fertnstert.2005.12.018. PMID 16759928
- [Background] Lim KJ, Odukoya OA, Ajjan RA, Li TC, Weetman AP, Cooke ID. The role of T-helper cytokines in human reproduction. Fertil Steril. 2000 Jan;73(1):136-42. doi: 10.1016/s0015-0282(99)00457-4. PMID 10632428
- [Background] Faas M, Bouman A, Moesa H, Heineman MJ, de Leij L, Schuiling G. The immune response during the luteal phase of the ovarian cycle: a Th2-type response? Fertil Steril. 2000 Nov;74(5):1008-13. doi: 10.1016/s0015-0282(00)01553-3. PMID 11056250
- [Background] Rier SE. Environmental immune disruption: a comorbidity factor for reproduction? Fertil Steril. 2008 Feb;89(2 Suppl):e103-8. doi: 10.1016/j.fertnstert.2007.12.040. PMID 18308048
- See also: The luteal phase after 3 decades of IVF: what do we know? HM Fatemi, Vol.19 Suppl. 4, 2009 Reproductive BioMedicine Online — http://www.rbmonline.com